CLINICAL TRIAL: NCT06542068
Title: Effectiveness of Using Chatbots for Nursing Students to Improve Mental Health and Reduce Stress During Internships.
Brief Title: Chatbot Effectiveness for Improving Mental Health and Reducing Stress in Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Kuo Ya-Wen, professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 113-470
Record Dates: First submitted 2024-07-29; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Mental Health; Stress; Nursing Education
Keywords: Internship Support; Chatbot Assistance; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Line Bot Assistance Group (Experimental): During the internship, students will use the Line Bot as a support tool.The Line Bot aims to provide psychological health support and stress management resources, helping students cope with stress and challenges encountered during their clinical internships.
  Interventions: Behavioral: Line Bot Assistance
- Control Group (No Intervention): This group will not receive assistance from the Line Bot chatbot. These students will receive only the regular internship support and resources without the use of any technological assistance tools.

INTERVENTIONS:
Behavioral: Line Bot Assistance — The chatbot is expected to provide self-help solutions and multiple counseling resources for stress and distress, options for face-to-face or online call requests, and a survey on mental health and stress.
  In terms of keywords, it will establish counseling response resources and methods for finding resources for special sensitive situations (e.g., feeling moody, suicidal, stressed, not wanting to intern, etc.).
  Arms: Line Bot Assistance Group

SUMMARY:
This study aims to evaluate the effectiveness of using a chatbot to improve mental health and reduce stress among nursing students during their internships. The study will be conducted through convenient sampling of nursing students from a technology university in southern Taiwan. Students will be divided into experimental and control groups to compare differences in mental health and stress levels after receiving support from the chatbot. Expected outcomes include gaining a better understanding of the fundamental characteristics of nursing students and their mental health and stress levels during internships. The results are expected to demonstrate that the chatbot can aid nursing students in handling typical internship issues, stress, and challenges, as well as in accessing mental health resources.

DETAILED DESCRIPTION:
Background: The number of suicides and the crude death rate among adolescents aged 15-24 have been gradually increasing. Nursing students experience greater stress compared to students from other disciplines, primarily due to the unfamiliar clinical environment, concerns about managing internships, and worries about their ability to accurately judge and handle patient conditions due to a lack of experience. The diverse and highly complex nature of clinical practice sites significantly impacts the mental health and stress levels of nursing students during their internships. Therefore, it is crucial to pay attention to the cultivation of nursing students as they enter clinical practice. In response to changing times, mobile devices and chatbot tools are critically important support resources for students.Objective:The aim is to understand how chatbot can help nursing students improve their mental health and stress during their internships. Methods:This study will employ a quasi-experimental design and will use convenience sampling to recruit nursing students from a technology university in southern Taiwan. Structured questionnaires will be used to collect data on basic demographic information, a brief health scale, and a clinical internship stress scale. It is estimated that 55 students will be recruited for both the experimental and control groups.Statistical analyses will be conducted using SPSS 28.0 software. Expected Outcomes: The expected outcomes of this study include gaining a better understanding of the basic attributes of nursing students and their mental health and stress levels during internships. The overall findings will serve as a reference for educational planning for nursing internship students and emphasize the importance of technology-assisted connections in practical learning within teaching policies.

ELIGIBILITY:
Inclusion Criteria:

Nursing students from the daytime four-year technical program at a university in southern Taiwan who have been scheduled for clinical internships.

Students who agree to participate in the study.

Exclusion Criteria:

Students who are only partially completing their internships (fragmented internship students).

Students who are unable to comply with the intervention measures.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-26 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Brief Symptom Rating Scale | The students are interning for four weeks. A pre-test was conducted during the first week, and a post-test was administered at the end of the fourth week.
  Five-point Likert-type scale of 0 to 4, with 0 being not at all and 4 being extremely.A total score on the BSRS-5 above 14, or a score of more than 1 on the additional suicide survey item, may indicate a severe mood disorder. Scores between 10 and 14 may indicate moderate mood disorders, and those between 6 and 9 could indicate mild mood disorders.
Clinical Internship Stress Survey Form | The students are interning for four weeks. A pre-test was conducted during the first week, and a post-test was administered at the end of the fourth week.
  Total of 24 questions are included in the survey, utilizing a four-point Likert-type scale ranging from 1 to 4. The total score on the scale falls between 24 and 96, with higher scores indicating increased stress levels during the clinical practicum.